CLINICAL TRIAL: NCT07125443
Title: Effect of Intraoperative Inhaled Nitric Oxide on Reperfusion Syndrome and Vasoplegia in Adult Liver Transplant Recipients: A Prospective Before-After Study
Brief Title: Effect Inhaled Nitric Oxide in Adult Liver Transplant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Raffael Zamper, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iNO for LT
Record Dates: First submitted 2025-08-07; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Liver Diseases; Reperfusion Injury; Vasoplegia
Keywords: Inhaled Nitric Oxide; Anesthesia
MeSH Terms: conditions — Liver Diseases; Reperfusion Injury; Vasoplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention Retrospective "Before" Group (Active Comparator): Adult liver transplant recipients identified retrospectively from the institutional transplant database, including all patients who underwent orthotopic liver transplantation since the implementation of the OneChart electronic medical record (EMR) system between the time period of January 1, 2020 - May 31, 2025.
  Interventions: Other: No Intervention Retrospective "Before" Group
- Prospective iNO Administration ("After" Group) (Experimental): Adult patients undergoing liver transplantation with prospective intervention involving intraoperative administration of inhaled nitric oxide (iNO) and prospective data collection.
  Interventions: Drug: Prospective iNO Administration ("After" Group)

INTERVENTIONS:
Drug: Prospective iNO Administration ("After" Group) — Adult patients undergoing liver transplantation after the implementation of the iNO protocol, with prospective intervention involving intraoperative administration of iNO and prospective data collection. Inhaled nitric oxide will be administered via the anesthesia machine, under the supervision of the attending Anesthesiologist, at a concentration of 20 parts per million (ppm) starting at induction of anesthesia. At the onset of the anhepatic phase (i.e., after explantation of the native liver), the concentration will be increased to 80 ppm. Administration will be continued until the end of the surgical procedure, at which point iNO will be discontinued.
  Arms: Prospective iNO Administration ("After" Group)
Other: No Intervention Retrospective "Before" Group — Adult liver transplant recipients identified retrospectively from the institutional transplant database, including all patients who underwent orthotopic liver transplantation since the implementation of the OneChart electronic medical record (EMR) system between the time period of January 1, 2020 - May 31, 2025.
  Arms: No Intervention Retrospective "Before" Group

SUMMARY:
Liver transplantation remains the only cure for patients with end-stage liver disease. Despite continuous advances in medical care, ischemia-reperfusion injury (IRI) (tissue damage that occurs when blood supply is restored to an area that has been deprived of oxygen) remains a major contributor to complications with the newly transplanted liver. IRI can lead to a condition known as post-reperfusion syndrome that involves profound narrowing of blood vessels, significantly low blood pressure, and an increased requirement of medication to control blood pressure. In some cases, post-reperfusion syndrome can progress to a condition known as post-reperfusion vasoplegia which is a condition where severely low blood pressure persists even after blood flow is restored to the liver. This is often accompanied by complications such as improperly functioning kidneys, blood clotting disorders, and complications with the transplanted liver that can significantly affect patient outcomes. Recent studies have shown than inhaled nitric oxide (a gas that can relax blood vessels) can reduce the severity of IRI in the liver. This study is being conducted to determine whether the administration of inhaled nitric oxide during surgery reduces the severity of post-reperfusion syndrome and the incidence of post-reperfusion vasoplegia in adult patients undergoing liver transplantation. This is a before-and-after study design that will involve both the retrospective collection of data between the time period of January 1, 2020 - May 31, 2025 and prospective interventions involving adult liver transplant recipients.

DETAILED DESCRIPTION:
Orthotopic liver transplantation remains the only curative option for patients with end-stage liver disease. Despite continuous advances in surgical techniques and perioperative management, ischemia-reperfusion injury (IRI) remains a major contributor to early graft dysfunction, with clinical consequences including prolonged intensive care stay, increased morbidity, and higher resource utilization. Reperfusion of the donor liver, particularly after portal and arterial unclamping, frequently triggers a hemodynamic instability known as post-reperfusion syndrome. This syndrome is characterized by profound vasodilation, hypotension, and a significant increase in vasopressor requirements. In some patients, it progresses into post-reperfusion vasoplegia, a state of sustained low systemic vascular resistance and poor end-organ perfusion. This condition is often accompanied by renal dysfunction, coagulopathy, and impaired early graft function, which significantly affect patient outcomes.

The pathophysiology of hepatic IRI is complex, involving endothelial activation, neutrophil recruitment, oxidative stress, mitochondrial dysfunction, and cytokine release. A key mechanistic factor contributing to reperfusion injury is the reduced bioavailability of nitric oxide (NO), due either to decreased production by endothelial nitric oxide synthase (eNOS) or its rapid inactivation by reactive oxygen species and heme-containing proteins. NO plays an essential role in maintaining microvascular tone, limiting leukocyte adhesion, and protecting against mitochondrial and endothelial injury. Restoration of NO signaling has been shown to protect against IRI in preclinical models. Inhaled nitric oxide (iNO) is approved for pulmonary hypertension and neonatal hypoxemia, but accumulating evidence suggests that it may also exert extrapulmonary effects. Studies in both animals and humans have demonstrated that iNO can attenuate IRI in the liver, heart, and skeletal muscle by increasing circulating nitrite and other bioactive NO metabolites that act as reservoirs and mediators of NO activity during ischemic stress.

In the context of liver transplantation, two retrospective clinical studies have shown that intraoperative iNO administration (at 80 ppm (parts per million)) is safe and may accelerate the recovery of liver function, reduce hepatocellular apoptosis, and decrease postoperative complications. These findings suggest that iNO could modulate the hemodynamic response to reperfusion and improve graft performance. However, despite these promising results, no prospective controlled trials or before-after studies have yet evaluated the real-time impact of intraoperative iNO on reperfusion syndrome and vasoplegia in liver transplantation.

The investigators hypothesize that the intraoperative administration of inhaled nitric oxide reduces the severity of reperfusion syndrome and the incidence of post-reperfusion vasoplegia in adult patients undergoing liver transplantation. Furthermore, the investigators propose that this intervention contributes to improved early graft function, particularly with regard to excretory performance. The present study aims to prospectively assess these outcomes using a before-after design, comparing matched cohorts of patients undergoing liver transplantation with and without intraoperative iNO. By addressing this existing gap in the literature, the investigators hope to generate clinically relevant data that may support the integration of iNO into standard perioperative protocols for liver transplant recipients.

This study involves 2 patient groups:

1. Retrospective "before" group (control arm): Adult liver transplant recipients identified retrospectively from the institutional transplant database, including all patients who underwent orthotopic liver transplantation since the implementation of the OneChart electronic medical record (EMR) system at London Health Sciences Centre between the time period of January 1, 2020 - May 31, 2025.
2. Prospective "after" group (intervention arm): 60 consecutive adult patients undergoing liver transplantation after the implementation of the iNO protocol, with prospective intervention involving intraoperative administration of iNO and prospective data collection.

For the prospective, "after" study group, the participant's liver transplant procedure will proceed according to plan. Informed, written consent will be obtained prior to the start of surgery.

Inhaled nitric oxide will be administered via the anesthesia machine, under the supervision of the attending Anesthesiologist, at a concentration of 20 parts per million (ppm) starting at induction of anesthesia. At the onset of the anhepatic phase (i.e., after explantation of the native liver), the concentration will be increased to 80 ppm. Administration will be continued until the end of the surgical procedure, at which point iNO will be discontinued. Standard anesthesia and transplant protocols will be followed in both groups, with no additional changes aside from the administration of iNO.

Participation in the "before" group will only involve retrospective data collection from the patients' electronic medical record that will gather data collected during the period of January 1, 2020 - May 31, 2025.

Data that will be collected include demographic data, medical history, intraoperative surgical details, details of iNO administration (where applicable), and post-operative outcomes. The timeline for collecting postoperative outcomes will be between 0-72 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Undergoing or underwent (for the retrospective "before" group) primary orthotopic liver transplantation. Retrospective data collection for retrospective group will take place between January 1, 2020 - May 31, 2025.
* Written informed consent obtained for patients in the prospective ("after") group

Exclusion Criteria:

* History of pulmonary arterial hypertension (mean pulmonary artery pressure ≥ 25 mmHg)
* Re-transplantation
* Acute fulminant hepatitis
* Combined organ transplantation (e.g., liver-kidney)
* Lack of complete data for propensity matching - Inability to communicate in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Impact of nitric oxide to reduce the severity of post-reperfusion syndrome in adult patients undergoing liver transplantation | 0-72 hours following liver transplant
  This will be measured by considering the following parameters for these indications following iNO administration:
  • Incidence of post-reperfusion syndrome, defined as a ≥30% drop in mean arterial pressure within 5 minutes of reperfusion, lasting for more than 1 minute
Impact of nitric oxide to reduce the incidence of incidence of post-reperfusion vasoplegia in adult patients undergoing liver transplantation | 0-72 hours following liver transplant
  This will be measured by considering the following parameters for these indications following iNO administration:
  • Incidence of vasoplegia, defined as persistent hypotension requiring norepinephrine ≥ 0.1 µg/kg/min for ≥ 30 minutes despite adequate volume resuscitation

SECONDARY OUTCOMES:
Impact of intraoperative administration of inhaled nitric oxide (iNO) on patient hospital stay. | 0-72 hours following liver transplant
  This will be measured by evaluating:
  • Length of ICU and hospital stay (measured in days).
Impact of intraoperative administration of inhaled nitric oxide (iNO) on in-hospital mortality | 0-72 hours following liver transplant
  This will be measured by evaluating:
  -In-hospital mortality
Impact of intraoperative administration of inhaled nitric oxide (iNO) on liver function | 0-72 hours following liver transplant
  This will be measured by evaluating:
  - Peak serum ALT (Alanine Aminotransferase) and AST (Aspartate Aminotransferase) levels (measured in international units per litre (U/L)
Impact of intraoperative administration of inhaled nitric oxide (iNO) on blood clotting | 0-72 hours following liver transplant
  This will be measured by evaluating the following:
  - Time to INR (International Normalized Ratio) normalization
Impact of intraoperative administration of inhaled nitric oxide (iNO) on early graft dysfunction | 0-72 hours following liver transplant
  This will be measured by the Olthoff criteria
Impact of intraoperative administration of inhaled nitric oxide (iNO) on the requirements for post-operative therapies and medications. | 0-72 hours following liver transplant
  This will be measured by recording the need for patients to receive the following after surgery:
  * Postoperative vasopressor requirement
  * Renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Raffael Zamper, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang JD Jr, Smith AB, Brandon A, Bradley KM, Liu Y, Li W, Crowe DR, Jhala NC, Cross RC, Frenette L, Martay K, Vater YL, Vitin AA, Dembo GA, Dubay DA, Bynon JS, Szychowski JM, Reyes JD, Halldorson JB, Rayhill SC, Dick AA, Bakthavatsalam R, Brandenberger J, Broeckel-Elrod JA, Sissons-Ross L, Jordan T, Chen LY, Siriussawakul A, Eckhoff DE, Patel RP. A randomized clinical trial testing the anti-inflammatory effects of preemptive inhaled nitric oxide in human liver transplantation. PLoS One. 2014 Feb 12;9(2):e86053. doi: 10.1371/journal.pone.0086053. eCollection 2014. PMID 24533048
- [Background] Lang JD Jr, Teng X, Chumley P, Crawford JH, Isbell TS, Chacko BK, Liu Y, Jhala N, Crowe DR, Smith AB, Cross RC, Frenette L, Kelley EE, Wilhite DW, Hall CR, Page GP, Fallon MB, Bynon JS, Eckhoff DE, Patel RP. Inhaled NO accelerates restoration of liver function in adults following orthotopic liver transplantation. J Clin Invest. 2007 Sep;117(9):2583-91. doi: 10.1172/JCI31892. PMID 17717604
- [Background] Jaeschke H. Reactive oxygen and mechanisms of inflammatory liver injury. J Gastroenterol Hepatol. 2000 Jul;15(7):718-24. doi: 10.1046/j.1440-1746.2000.02207.x. PMID 10937675
- [Background] Kubes P, Suzuki M, Granger DN. Nitric oxide: an endogenous modulator of leukocyte adhesion. Proc Natl Acad Sci U S A. 1991 Jun 1;88(11):4651-5. doi: 10.1073/pnas.88.11.4651. PMID 1675786
- [Background] Bataller R, Brenner DA. Liver fibrosis. J Clin Invest. 2005 Feb;115(2):209-18. doi: 10.1172/JCI24282. PMID 15690074
- [Background] Duranski MR, Greer JJ, Dejam A, Jaganmohan S, Hogg N, Langston W, Patel RP, Yet SF, Wang X, Kevil CG, Gladwin MT, Lefer DJ. Cytoprotective effects of nitrite during in vivo ischemia-reperfusion of the heart and liver. J Clin Invest. 2005 May;115(5):1232-40. doi: 10.1172/JCI22493. Epub 2005 Apr 14. PMID 15841216
- [Background] Cannon RO 3rd. Role of nitric oxide in cardiovascular disease: focus on the endothelium. Clin Chem. 1998 Aug;44(8 Pt 2):1809-19. PMID 9702990